CLINICAL TRIAL: NCT00528385
Title: Influence of Adding Aldosterone Receptor Blocker to Dual Renin-Angiotensin-Aldosterone System Blockade on Proteinuria
Brief Title: Optimalization of Nephroprotection Using Agents Inhibiting Renin-Angiotensin-Aldosterone System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ST-4/RAAS/02
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2007-09-12 (Estimated); Status verified 2007-09

CONDITIONS: Chronic Kidney Disease; Proteinuria
Keywords: Proteinuria; Renin-Angiotensin-Aldosterone System; Aldosterone Antagonists
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Spironolactone; Canrenoic Acid

INTERVENTIONS:
Drug: Spironolactone (Spironol) 25 mg — In the 8-weeks run-in period ACEI, cilazapril (5 mg), telmisartan (80 mg) and hydrochlorotiazyd (12.5 mg) were administered to achieve the target blood pressure below 130/80 mmHg. Next, they were randomly assigned to add (or not) 25 mg of spironolactone in two active treatment periods lasting 8 weeks each.

SUMMARY:
The main purpose of the study is find whether the addition of aldosterone antagonist, spironolactone to dual renin-angiotensin-aldosterone system blockade involving angiotensin converting enzyme inhibitor and AT-1 angiotensin II receptor blocker leads to the reduction of proteinuria, main prognostic marker of chronic kidney disease progression.

DETAILED DESCRIPTION:
The renin-angiotensin-aldosterone system (RAAS) plays an important role in the progression of chronic kidney diseases (CKD), and inhibition of the RAAS with angiotensin-converting enzyme inhibitors (ACEI) and angiotensin II type 1 receptor blockers (ARB) may retard CKD progression. Dual pharmacological blockade of the RAAS with ACEI and ARB is recommended as a standard renoprotective management at least in patients with nondiabetic proteinuric CKD. However, neither ACEI nor ARB, even in high doses or in concomitant usage, abrogate the progression of CKD completely. Innovative approaches are needed to keep patients with CKD off dialysis. Additional blockade of the aldosterone pathway may prove to be such beneficial therapeutic concept.Aldosterone, a final effector of RAAS plays a significant role in the pathogenesis of CKD independently of angiotensin II through direct cellular action. This includes promoting an inflammatory response, endothelial dysfunction, and fibrosis by increasing plasminogen activator inhibitor (PAI-1) and transforming growth factor beta-1 (TGF-beta-1) expression and stimulation reactive oxygen species.A number of observations suggest nongenomic vasoconstrictor action of aldosterone leading to raise arterial and glomerular capillary pressure.Given these facts additional administration of aldosterone antagonist to combination treatment with ACEI and ARB, so called triple RAAS blockade may provide additional renal protection. To shed more light on this issue, we performed a randomised open controlled study to evaluate the influence of triple RAAS therapy on surrogate markers of kidney injury, i.e. proteinuria, markers of tubular involvement and kidney fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease
* stable proteinuria above 300 mg/24 hours (no variations above 25% in the last 6 months)
* normal or slightly impaired stable renal function defined as serum creatinine level below 1.7 mg/dl (eGFR > 45 ml/min)

Exclusion Criteria:

* nephrotic syndrome
* steroids or other immunosuppressive treatment minimum during six months before the study
* diabetes mellitus
* potassium serum level > 5.1 mEq/L
* albumin serum level < 2.0mg/dL
* creatinine serum level >2 mg/dl
* current diagnosis of heart failure New York Heart Association (NYHA) Class II-IV
* clinically significant valvular heart disease or second or third degree heart block without a pacemaker
* history of hypertensive encephalopathy, cerebrovascular accident or transient ischemic cerebral attack
* history of myocardial infarction, unstable angina pectoris, coronary bypass surgery, or any percutaneous coronary intervention
* history of malignancy including leukemia and lymphoma (but not basal cell skin carcinoma) within the past five years
* pregnant or nursing women
* any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs.
* history of alcohol abuse
* NSAID abuse (more than 2 doses per week)
* known or suspected contraindications to the study medications, including history of allergy to ACE inhibitors, AT-1 receptor blockers and aldosterone antagonists

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2005-03

PRIMARY OUTCOMES:
Investigate the antiproteinuric effect of adding aldosterone antagonist, spironolactone to the combination therapy with angiotensin converting enzyme inhibitor and AT-1 receptor blocker in maximal recommended doses.

SECONDARY OUTCOMES:
Investigate the effect of the study intervention on urine excretion of N-acetyl-β-D-glucosaminidase, alfa1-microglobulin and amino-terminal propeptide of type III procollagen.

CONTACTS AND LOCATIONS:
Overall Officials: Boleslaw Rutkowski, MD, PhD, Principal Investigator — Department of Nephrology Transplantology and Internal Medicine. Medical University of Gdansk.

REFERENCES:
- [Derived] Cooper TE, Teng C, Tunnicliffe DJ, Cashmore BA, Strippoli GF. Angiotensin-converting enzyme inhibitors and angiotensin receptor blockers for adults with early (stage 1 to 3) non-diabetic chronic kidney disease. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD007751. doi: 10.1002/14651858.CD007751.pub3. PMID 37466151
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592